CLINICAL TRIAL: NCT02419872
Title: A Phase IV Real-World Multi-Country Observational Study on Patients' Disease Control and Self-Reported Outcomes During Fixed Dose Combination Inhaler Treatment for Persistent Asthma and COPD
Brief Title: Study in Patients' With Persistent Asthma and Chronic Obstructive Pulmonary Disease
Acronym: SPRINT
Status: Completed | Type: Observational
Sponsor: Teva Pharmaceuticals Europe (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: BFS-AS-40087
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Participants: Patients are confirmed to have either Persistent Asthma or COPD
  Interventions: Drug: Marketed antagonists

INTERVENTIONS:
Drug: Marketed antagonists — Medication for each patient is determined by the physician based on the patient's individual clinical profile and in accordance with the approved indication and label of the prescribed drug
  Other Names: as prescribed

SUMMARY:
The study is to evaluate the percentage of patients with asthma or COPD achieving disease control

DETAILED DESCRIPTION:
There are no treatment groups or interventions to which the patients can be randomly assigned. Data will be collected in a routine setting on a single occasion during an otherwise normal visit at the physician's office or clinic. Participating physicians will not perform any medical procedures that are outside of their normal daily clinical practice. All treatment decisions are at the sole discretion of the participating physicians and reflect their current standard of care

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age who has been diagnosed with persistent asthma or patient ≥ 40 years of age and/or (ex)-smoker with more than 10 pack years of smoking who has been diagnosed with COPD
* Treatment with a stable dose (no change in dose or change by less than 50% in the last 3 months) of a Inhaled corticosteroid (ICS), Long-acting beta2-agonists (LABA), Fixed dose combination (FDC) administered twice daily by Dry powder inhaler (DPI) for 3 months prior to enrollment in accordance with its approved indication
* Patient is willing and able to provide written informed consent;
* Patient agrees to participate in the study and to disclose any medical events to the treating physician;
* Patient is able to complete the questionnaires.

Exclusion Criteria:

• Current enrolment or planned enrolment in an interventional study (patients are allowed to participate in other observational or case-control studies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with asthma or COPD and on a stable dose of Inhaled corticosteroid (ICS)/Long-acting beta2-agonists (LABA) Fixed dose combination (FDC) administered by dry powder inhaler (DPI) twice daily for the previous 3 months
Sampling Method: Non-Probability Sample
Enrollment: 1743 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose respiratory disease is well controlled | 1 Day
  Questionnaires capture descriptive, qualitative responses

SECONDARY OUTCOMES:
Patient Satisfaction Score | 1 Day
  A 10-point scale (where 1 = "not at all satisfied" and 10 = "extremely satisfied") is used to assess the patients' satisfaction
Proportion of patients who comply with treatment according to Morisky Medication Adherence Scale (MMAS-8) | 1 Day
  The 8-item MMAS-8 is a self-reported instrument to measure medication adherence
Most Important Inhaler Features (MIIF) questionnaire | 1 Day
  MIIF is a 10-point rating scale (where 1 = "not at all easy" and 10 = "extremely easy") for the 5 most important features
Percentage of Participants with Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals USA
Locations (141):
- Croatia (13):
  - Teva Investigational Site 1011, Dubrovnik
  - Teva Investigational Site 1001, Karlovac
  - Teva Investigational Site 1007, Karlovac
  - Teva Investigational Site 1015, Metković
  - Teva Investigational Site 1014, Pula
  - Teva Investigational Site 1012, Rijeka
  - Teva Investigational Site 1005, Samobor
  - Teva Investigational Site 1004, Sisak
  - Teva Investigational Site 1013, Varaždin
  - Teva Investigational Site 1006, Zadar
  - Teva Investigational Site 1002, Zagreb
  - Teva Investigational Site 1003, Zagreb
  - Teva Investigational Site 1008, Zagreb
- Denmark (7):
  - Teva Investigational Site 201, Aalborg
  - Teva Investigational Site 202, Aarhus
  - Teva Investigational Site 207, Copenhagen
  - Teva Investigational Site 204, Hvidovre
  - Teva Investigational Site 205, Kolding
  - Teva Investigational Site 203, Næstved
  - Teva Investigational Site 206, Roskilde
- Ireland (6):
  - Teva Investigational Site 905, Enniscorthy
  - Teva Investigational Site 904, Lifford
  - Teva Investigational Site 903, Mallow
  - Teva Investigational Site 901, Sligo
  - Teva Investigational Site 906, Tramore
  - Teva Investigational Site 902, Youghal
- Italy (29):
  - Teva Investigational Site 513, Ancona
  - Teva Investigational Site 31, Bari
  - Teva Investigational Site 512, Brescia
  - Teva Investigational Site 502, Brindisi
  - Teva Investigational Site 514, Catania
  - Teva Investigational Site 9, Chieti
  - Teva Investigational Site 22, Florence
  - Teva Investigational Site 505, Foggia
  - Teva Investigational Site 20, Genova
  - Teva Investigational Site 30, Lecco
  - Teva Investigational Site 509, Legnago
  - Teva Investigational Site 3, Modena
  - Teva Investigational Site 11, Napoli
  - Teva Investigational Site 8, Napoli
  - Teva Investigational Site 14, Orbassano
  - Teva Investigational Site 508, Palermo
  - Teva Investigational Site 516, Parma
  - Teva Investigational Site 501, Pavia
  - Teva Investigational Site 10, Perugia
  - Teva Investigational Site 18, Pietra Ligure
  - Teva Investigational Site 506, Pisa
  - Teva Investigational Site 510, Pordenone
  - Teva Investigational Site 503, Roma
  - Teva Investigational Site 21, Sassari
  - Teva Investigational Site 24, Scafati
  - Teva Investigational Site 515, Sesto San Giovanni
  - Teva Investigational Site 507, Siena
  - Teva Investigational Site 4, Torino
  - Teva Investigational Site 511, Verona
- Netherlands (7):
  - Teva Investigational Site 606, Alkmaar
  - Teva Investigational Site 604, Grubbenvorst
  - Teva Investigational Site 601, Harderwijk
  - Teva Investigational Site 602, Helmond
  - Teva Investigational Site 607, Hoofddorp
  - Teva Investigational Site 603, Hoorn
  - Teva Investigational Site 605, Rotterdam
- Norway (4):
  - Teva Investigational Site 302, Hamar
  - Teva Investigational Site 303, Holter
  - Teva Investigational Site 301, Oslo
  - Teva Investigational Site 304, Oslo
- Portugal (7):
  - Teva Investigational Site 702, Aveiro
  - Teva Investigational Site 707, Barcelos
  - Teva Investigational Site 706, Braga
  - Teva Investigational Site 701, Covilha
  - Teva Investigational Site 703, Guimarães
  - Teva Investigational Site 705, Porto
  - Teva Investigational Site 704, Vila Nova de Gaia
- Spain (43):
  - Teva Investigational Site 119, A Coruña
  - Teva Investigational Site ES044, A Coruña
  - Teva Investigational Site 113, Alcorcón
  - Teva Investigational Site ES048, Alcorcón
  - Teva Investigational Site 101, Barcelona
  - Teva Investigational Site 102, Barcelona
  - Teva Investigational Site 132, Barcelona
  - Teva Investigational Site 133, Cáceres
  - Teva Investigational Site 114, Córdoba
  - Teva Investigational Site 111, Jaén
  - Teva Investigational Site 105, Laredo
  - Teva Investigational Site 120, Lugo
  - Teva Investigational Site 109, Madrid
  - Teva Investigational Site 110, Madrid
  - Teva Investigational Site 124, Madrid
  - Teva Investigational Site 126, Madrid
  - Teva Investigational Site 134, Madrid
  - Teva Investigational Site 136, Madrid
  - Teva Investigational Site 135, Manacor
  - Teva Investigational Site 108, Málaga
  - Teva Investigational Site 118, Málaga
  - Teva Investigational Site 123, Málaga
  - Teva Investigational Site ES049, Málaga
  - Teva Investigational Site 128, Murcia
  - Teva Investigational Site 103, Oviedo
  - Teva Investigational Site 107, Pamplona
  - Teva Investigational Site 130, Ponferrada
  - Teva Investigational Site 131, Pontevedra
  - Teva Investigational Site 139, Santa Cruz de Tenerife
  - Teva Investigational Site 117, Santander
  - Teva Investigational Site 106, Santiago de Compostela
  - Teva Investigational Site 112, Seville
  - Teva Investigational Site 122, Seville
  - Teva Investigational Site 125, Seville
  - Teva Investigational Site ES046, Seville
  - Teva Investigational Site 129, Terrassa
  - Teva Investigational Site 140, Teruel
  - Teva Investigational Site 104, Valencia
  - Teva Investigational Site 115, Valencia
  - Teva Investigational Site 116, Valencia
  - Teva Investigational Site 127, Valencia
  - Teva Investigational Site 121, Vic
  - Teva Investigational Site 138, Zaragoza
- Teva Investigational Site 401, Lund, Sweden
- United Kingdom (24):
  - Teva Investigational Site 804, Atherstone
  - Teva Investigational Site 803, Beccles
  - Teva Investigational Site 813, Belfast
  - Teva Investigational Site 816, Birkenhead
  - Teva Investigational Site 815, Bolton
  - Teva Investigational Site 812, Bridgwater
  - Teva Investigational Site 807, Chippenham
  - Teva Investigational Site 817, Doncaster
  - Teva Investigational Site 811, Hinckley
  - Teva Investigational Site 801, Hitchin
  - Teva Investigational Site 821, Nantwich
  - Teva Investigational Site 824, Norwich
  - Teva Investigational Site 806, Portsmouth
  - Teva Investigational Site 808, Royal Leamington Spa
  - Teva Investigational Site 820, Sandbach
  - Teva Investigational Site 805, Thaxted
  - Teva Investigational Site 818, Thornton-Cleveleys
  - Teva Investigational Site 819, Tollerton
  - Teva Investigational Site 809, Trowbridge
  - Teva Investigational Site 802, Watford
  - Teva Investigational Site 822, Wells-next-the-Sea
  - Teva Investigational Site 810, Winchester
  - Teva Investigational Site 814, Wolverhampton
  - Teva Investigational Site 823, Wymondham